CLINICAL TRIAL: NCT02085330
Title: Hyperbaric Oxygen Therapy in Patients Suffering From Mild Cognitive Impairment and Vascular Subcortical Ischemia
Brief Title: Hyperbaric Oxygen Therapy for Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Dr. Shai Efrati, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 69/13
Record Dates: First submitted 2014-03-11; First posted 2014-03-12 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Mild Cognitive Impairment and Vascular Subcortical Ischemia
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyperbaric oxygen therapy (Experimental): Hyperbaric oxygen therapy
  Interventions: Device: Hyperbaric oxygen therapy
- Standard follow up (No Intervention)

INTERVENTIONS:
Device: Hyperbaric oxygen therapy — 100%, 2 ATA, 90 minutes
  Arms: Hyperbaric oxygen therapy

SUMMARY:
Dementia is a very frequent cognitive disorder among elderly individuals. Its prevalence is about 15-20% of the population over the age of 65. The most common forms of dementia among the elderly demented patients are Alzheimer's disease (AD) (prevalence of 70%) and Vascular dementia (VD) (prevalence of about 30-40%).There is also a high rate (about 40%) of coexisting of AD and VD among the dementia patients, defined as mixed dementia.

Mild Cognitive Impairment (MCI) is a pre-dementia phase of cognitive decline. It is also considered as a prodromal phase of both VD and AD. Its basic clinical features include: cognitive concern, reflecting a change in cognition, reported by the patient or informant (i.e., historical or observed evidence of decline over time), with objective evidence of impairment in one or more cognitive domains (i.e., by formal cognitive testing), as well as preservation of independence in functional abilities and not being demented (i.e., no significant impairment social or occupational functioning).

Hyperbaric oxygen therapy (HBOT) has been investigated for treatment of numerous diseases for more than 300 years. The principal effect of HBOT is increasing the solubility of oxygen in plasma to a level sufficient to support tissues with minimal oxygen supply carried on by hemoglobin. Clinical studies published this year present convincing evidence that hyperbaric oxygen therapy (HBOT) can be the coveted neurotherapeutic method for brain repair. Thus, it seems that HBOT might be an efficient and clinically feasible method capable of increasing tissue/cellular oxygenation and effectively evoking neuroplasticity in the chronically vascular-lesioned areas during the post microvascular lesion phase.

This is a prospective, randomized, control crossed over, study evaluating the effect of HBOT in patients suffering from Mild Cognitive Impairment and Vascular Subcortical Ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as suffering from Mild Cognitive Impairment by-National Institute on Aging Alzheimer Association criteria.
* Patients diagnosed as suffering from MCI to be due to Vascular Subcortical Ischemia by subcortical vascular changes in MRI, according to the MRI protocol of the European multicenter leukoaraiosis and disability study protocol.
* At least 1 of the following vascular risk factors arterial hypertension or known hypertension treated by blood pressure lowering medications, hypercholesterolemia.
* The onset of the disease is slow and gradual
* The course is continuously or step-like progressive for more than 1 year
* Patients who are ambulatory
* No other active neurological, systemic or psychiatric conditions that might be the primary cause of the current syndrome or significantly affect the current cognitive disorder.
* No previous brain disorder except the current contingency of the cognitive disorder.
* Balanced systemic psychiatric state for the past 3 months.

Exclusion Criteria:

* Dynamic neurologic improvement or worsening during the last month
* Had been treated with HBOT for any other reason prior to their inclusion
* Have any other indication for HBOT
* Chest pathology incompatible with pressure changes
* Inner ear disease
* Patients suffering from claustrophobia
* Patients suffering from any active malignant disease
* Inability to sign written informed consent.
* Patients with cognitive changes which cannot be defined as Mild Cognitive Impairment by National Institute on Aging Alzheimer Association criteria and global CDR score.
* Patients who do not have Vascular Subcortical Ischemia by the subcortical vascular changes in MRI according to the European multicenter leukoaraiosis and disability study protocol.
* The onset of the disease is not slow and gradual.
* The course is not continuously or step like progressive for more than 1 year.
* Patients who are not ambulatory
* There are other active neurological, systemic or psychiatric conditions that might be the primary cause of the current syndrome or significantly affect the current cognitive disorder.
* Any previous brain disorder except the current contingency of the cognitive disorder.
* Patients whose systemic psychiatric state is not balanced for the past 3 months.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-05 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Vascular Dementia Assessment Scale cognitive subscale (VADAS-cog) | 3 months

SECONDARY OUTCOMES:
Daily functioning, autonomy and quality of life | 3 months
Safety of HBOT in patients with mci | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel